CLINICAL TRIAL: NCT04335955
Title: Platelet Indices in Prediction of Mortality in Critically Ill Septic Patients
Status: Completed | Type: Observational
Sponsor: Amany Faheem (Other)
Responsible Party: Sponsor-Investigator, Amany Faheem, sponsor investigator, Tanta University
Organization: Tanta University (Other)
Other Study IDs: Platelet Indices in sepsis
Record Dates: First submitted 2020-04-03; First posted 2020-04-07 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Platelet Indices; Mortality; Sepsis
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Platelets (PLT), a major and essential constituent of blood, plays an important role in physiological and pathological processes such as coagulation, thrombosis, inflammation and maintenance of vascular endothelial cells the integrity (1).

Platelet indices are a group of parameters that are used to measure the total amount of PLTs, PLTs morphology and proliferation kinetics (2).

The commonly used PLT indices include PLT count, mean platelet volume (MPV), platelet distribution width (PDW), and plateletcrit (PCT). The MPV refers to the ratio of PCT to PLT count. PDW is numerically equal to the coefficient of PLT volume variation, which is used to describe the dispersion of PLTs volume (3).

It is well known that platelet indices have been applied in the diagnosis of hematological system diseases. In recent years, it has been discovered that these indices are related to the severity of illness and patients' prognosis. Reduction in PLT count is an independent risk factor for critically ill patients in intensive care unit (4).

In addition, Acute Physiology and Chronic Health Evaluation II (APACHE II) System also includes thrombocytopenia as an independent risk factor for mortality (5).

In a recent research, it will be reported that MPV will be rising with interleukin-6 and C-reactive protein in septic premature infants. MPV has been used as predictor of many inflammatory diseases as MPV significantly higher on both day 1 and day 3 in neonatal sepsis (6).

In addition, in patients with cirrhosis and ascites, elevated PDW and MPV will be accurate diagnostic predictors for ascetic fluid infection (7).

MPV and PDW will be used as biomarkers predicting the development of postoperative sepsis in colorectal cancer patient (8).

All these evidences indicated that PLT indices will be considered as indicator in a series of diseases (9).

Advantages of platelet indices are simple, available, cheap tools and routinely done in the hospital laboratory in all critical ill patients and may be a useful, sensitive tool for diagnosis and monitoring these patients especially in limited resource countries as Egypt. However, whether PLT indices are correlated with procalcitonin in assessment the severity of illness is still under research in septic patients

DETAILED DESCRIPTION:
Blood will be drawn from the peripheral vein, arterial or a central catheter for evaluation of whole blood count, C-reactive protein (CRP), and procalcitonin serum levels. This procedure will be done at diagnosis, 3, 7, 14, 21 and 28 days of sepsis.

The following data will be recorded:

* Demographic data (age, gender and BMI) and cause of sepsis
* Procalcitonin and its correlation with changes in platelet indices
* The odds ratio (OR) for mortality in patients with normal and abnormal platelet indices.
* Sequential organ failure assessment (SOFA) scores.

ELIGIBILITY:
Inclusion Criteria:

patients aged 18-65 years ICU stay more than 24 hours septic patients according to Third International Consensus Definitions Septic Shock patients according to Third International Consensus Definitions

Exclusion Criteria:

* Pregnant women
* Patients with active hemorrhage
* Patients with hematological diseases (including anemia, hypersplenism
* Lymphoma or leukemia
* Rheumatism, and bone marrow diseases)
* Patients who had infused with blood or platelets prior to their admission
* Patients who had used anti-platelet drugs prior to their admission
* Patients who had received radiotherapy or chemotherapy or bone marrow transplantation 1 month prior to admission.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sepsis: life-threatening organ dysfunction caused by a dysregulated host response to infection. According to the 2016 consensus definitions, an increase in SOFA score of 2 or more constitutes organ dysfunction
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
The correlation between platelet indices and 30 days mortality among critically ill septic patients | within 30 days from hospital admission
  The correlation between platelet indices and 30 days mortality among critically ill septic patients

SECONDARY OUTCOMES:
Correlation between platelet indices and Length of ICU stay (days) | within 30 days from hospital admission
  Correlation between platelet indices and Length of ICU stay (days)
Correlation between platelet indices and detection of organs dysfunction | within 30 days from hospital admission
  Correlation between platelet indices and detection of organs dysfunction
Correlation between platelet indices and procalcitonin. | within 30 days from hospital admission
  Correlation between platelet indices and procalcitonin.

CONTACTS AND LOCATIONS:
Locations (1):
- Amany Afheem, Tanta, Egypt